CLINICAL TRIAL: NCT05591079
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of CS0159 in the Treatment of Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of CS0159 in Subjects With NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NASH-CS0159-002
Record Dates: First submitted 2022-10-09; First posted 2022-10-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-07

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1.4mg CS0159 (Experimental): One tablet daily for 12 weeks
  Interventions: Drug: CS0159 (Linafexor)
- 2mg CS0159 (Experimental): One tablet daily for 12 weeks
  Interventions: Drug: CS0159 (Linafexor)
- PLACEBO (Placebo Comparator): One tablet daily for 12 weeks
  Interventions: Drug: CS0159 (Linafexor)

INTERVENTIONS:
Drug: CS0159 (Linafexor) — Oral QD
  Other Names: placebo

SUMMARY:
A randomized, double-blind study to assess the safety, tolerability, PK and efficacy of CS0159 in subjects with Non-Alcoholic Steatohepatitis (NASH)

DETAILED DESCRIPTION:
This will be a multicenter, double-blind, randomized, placebo-controlled, dose-ranging study to evaluate the safety, tolerability, PKs, and efficacy of CS0159 in the treatment of patients with NASH over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnosis of NASH.
2. Evidence of metabolic syndrome, except for those patients with biopsy-proven NASH.
3. Body mass index (BMI) >25 kg/m2, NOTE: for Asian-Americans BMI >23 kg/m2.
4. Stable use of other antidiabetic, weight loss, or lipid-modifying medications for at least 12 weeks prior to randomization.

Exclusion Criteria:

1. Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days, whichever is longer.
2. Previous exposure to farnesoid X receptor (FXR) agonists 3 months prior to the first dosing.
3. Current or within 6 months of screening use of drugs associated with steatosis, including but not limited to eg, methotrexate, amiodarone, high-dose estrogen, tamoxifen, long term systemic steroids, anabolic steroids, valproic acid.
4. Prothrombin time international normalized ratio >1.3, unless due to therapeutic anticoagulation.
5. Total bilirubin >upper limit of normal (ULN; except for patients with Gilbert's syndrome with a normal direct bilirubin value and normal reticulocyte count).

   Platelet count <140 000/mm³, absolute neutrophil count <1500 cells/mm3, or total
6. white blood cells <3000 cells/mm3.
7. Alanine aminotransferase and aspartate aminotransferase (AST) >5 × ULN, or alkaline phosphatase (ALP) >1.5 × ULN.
8. Weight changes >10% in 6 months prior to screening, or weight changes >5% from the screening MRI-PDFF to randomization or from the time of the diagnostic liver biopsy to randomization, whichever is longer.
9. Poorly controlled hypertension (systolic >160 mm Hg, or diastolic blood pressure >100 mm Hg - mean of 3 measurements).
10. Uncontrolled diabetes mellitus (hemoglobin A1c >10.0% during screening).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
MRI-PDFF | Week 12
  To assess the changes in liver steatosis through magnetic resonance imaging (MRI) proton density fat fraction (PDFF) from baseline to Week 12
Adverse events | Week 12
  To evaluate the safety and tolerability of CS0159 in patients with NASH treated over 12 weeks

SECONDARY OUTCOMES:
Cmax | week 6, week 12
  maximum concentration (Cmax) from baseline to Week 12
tmax | week 6, week 12
  time to maximum plasma concentration (tmax) from baseline to Week 12
t1/2 | week 6, week 12
  half-life (t1/2) from baseline to Week 12
AUC | week 6, week 12
  accumulation ratio of area under the concentration-time curve (AUC) in plasma from baseline to Week 12
Pharmacodynamics (PD) | week 6, week 12
  Plasma concentrations and PD parameters of the biomarkers of FXR target engagement fibroblast growth factor 19 and 7α-hydroxy-4-cholesten-3-one (C4) from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Rong Deng, Study Director — Cascade Pharmaceuticals, Inc
Locations (17):
- United States (17):
  - National Research Institute - Gardena, Gardena, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research - Panorama City, Panorama City, California
  - Velocity Clinical Research - Santa Ana, Santa Ana, California
  - Ocala GI Research, Lady Lake, Florida
  - Florida Research Institute, Lakewood, Florida
  - San Marcus Research Clinic, Inc - Miami, Miami, Florida
  - Floridian Clinical Research, LLC - Miami Lakes, Miami Lakes, Florida
  - Gastroenterology Associates of Ocala, Ocala, Florida
  - Oracle Clinical Research, College Park, Georgia
  - Metropolitan Gastroenterology Associates - Westbank Office and Endoscopy, Marrero, Louisiana
  - Raja M. Din MD, PLLC - Gastroenterology & Hepatology, Greenbelt, Maryland
  - Lucas Research, Morehead City, North Carolina
  - Texas Liver Institute (TLI) - Austin, Austin, Texas
  - Pioneer Research Solutions Inc - Houston - Stancliff Rd, Houston, Texas
  - The Texas Liver Institute, Inc., San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No